CLINICAL TRIAL: NCT05577572
Title: The Effect of Supplementary Probiotic in the Dysbiosis of Gut Microbiota Caused by Second Line Bismuth Containing Quadruple Therapy in Helicobacter Pylori Eradication- A Multicentered, Randomized Double Blind Placebo-controlled Trial
Brief Title: Second Line Bismuth Containing Quadruple Therapy With Supplementary Probiotic
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: 201912191MIPC
Record Dates: First submitted 2021-06-14; First posted 2022-10-13 (Actual); Last update posted 2022-10-21 (Actual); Status verified 2022-09

CONDITIONS: H.Pylori Gastrointestinal Disease
Keywords: supplementary pylori; Bismuth quadruple therapy; H. pylori eradication

STUDY DESIGN:
Intervention Model Description: 200 patients are divided into two groups: one group receive probiotic for treatment period and the other group receive placebo. The treatment period is designed for 56 days: Bismuth containing quadruple therapy is performed from day 1~10 and probiotic (or placebo) is taken from day 1~56.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Probiotics packets (Experimental): Probiotics contains 450 billion colony-forming units per packet. The compositions are maltose, lactic acid bacteria and bifidobacteria blend, cornstarch, silicon dioxide.
  Interventions: Dietary Supplement: Probiotics packets
- Placebo packets (Placebo Comparator): The compositions are maltodextrin, silicon dioxide, sucralose
  Interventions: Dietary Supplement: Placebo packets

INTERVENTIONS:
Dietary Supplement: Probiotics packets — The treatment period is designed for 56 days: Bismuth containing quadruple therapy is performed from day 1~10 and Probiotics packets is taken from day 1~56.
  Arms: Probiotics packets
Dietary Supplement: Placebo packets — The treatment period is designed for 56 days: Bismuth containing quadruple therapy is performed from day 1~10 and Placebo packets is taken from day 1~56.
  Arms: Placebo packets

SUMMARY:
This study is designed to evaluate the clinical outcome of second line Bismuth containing quadruple therapy with supplementary probiotic for Helicobacter pylori eradication

DETAILED DESCRIPTION:
The role of Helicobacter pylori infection in the development of peptic ulcer disease and gastric cancer have been studied extensively. Eradication of H. pylori decreases the incidence of peptic ulcer and also gastric cancer. First line therapies for H. pylori eradication with PPI and antibiotic combinations considering local clarithromycin resistant rate reaching successful rates above 90%. Bismuth containing quadruple therapy (BQT), as a major choice of second line therapy, is widely prescribed but with considerable gastrointestinal side effects including diarrhea, nausea, vomiting, bloating and abdominal pain. Probiotics supplementation is defined as the adding of non-pathologic living microorgnisms. Numerous recent studies including meta-analyses and several randomized control trials revealed supplementary probiotics may improve the adverse effects and increase the successful rate of eradication therapy. Therefore, this study aim to assess the clinical impact of probiotics on Bismuth therapy and eradication of H. pylori.

It's a multicentered, randomized double blind placebo-controlled trial to evaluate the clinical outcome of second line Bismuth containing quadruple therapy with supplementary probiotic for Helicobacter pylori eradication. During the study, expected 200 patients failing in first-line Bismuth therapy would be enrolled in the trial. 200 patients are divided into two groups: one group receive probiotic for treatment period and the other group receive placebo. The treatment period is designed for 56 days: Bismuth containing quadruple therapy is performed from day 1~10 and probiotic (or placebo) is taken from day 1~56.

There are 5 visits for subjects to follow: day 0, day 10, day 56, 1 year and 3 years(optional). Esophagogastroduodenal scope for the pathology, H. pylori culture, susceptibility testing, genotypic resistance and virulence factors before D0. 13C-Urea breath tests are used to check Helicobacter pylori eradication on day 56, 1 year and 3 year. In addition to blood samples for general tests, stool samples would be collected on every visit to analyze gut microbiota.

ELIGIBILITY:
Inclusion Criteria:

Patients older than 20 years-old underwent documented non-Bismuth containing 1st line H. pylori eradication with failure defined by positive 13C-Urea Breath Test (13C-UBT) at least 6 weeks after completion of therapy is eligible to the study.

Exclusion Criteria:

1. History of gastrectomy, surgery in the small intestine or colon
2. History of gastric malignancy, including adenocarcinoma or lymphoma
3. Allergic history, history of severe adverse effects or contraindication to antibiotics (Tetracycline, Metronidazole ), proton pump inhibitor, or probiotics
4. Pregnant or lactating women
5. Severe concurrent chronic or acute disease (e.g. renal failure, liver cirrhosis, or active malignancy)
6. Concomitant use of clopidogrel or warfarin
7. Recent (<4 weeks) use of antibiotics, or recent (<4 weeks) probiotic use duration >2 weeks
8. Not able to give consent on blinding or randomizatio
9. Not able to give consent by his or herself

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2021-08-29 (Actual); Primary Completion 2023-04-29 (Estimated); Study Completion 2025-04-29 (Estimated)

PRIMARY OUTCOMES:
Evaluate the incidence of adverse effects after second line BQT between probiotic group (L) and placebo group (P) according to intentional to treat (ITT) and per-protocol (PP) analyses. | From Day 0 to Day 10.
  Adverse events are collected
Evaluate the incidence of adverse effects after second line BQT between probiotic group (L) and placebo group (P) according to intentional to treat (ITT) and per-protocol (PP) analyses. | From Day 0 to Day 56.
  Adverse events are collected

SECONDARY OUTCOMES:
Eradication rate of second line BQT between two groups | From Day 0 to Day 56.
  13C-Urea breath tests are performed to check the eradication of Helicobacter pylori between two groups
Dynamic changes in the gut microbiota between two groups | Day 0.
  Stool sample collection for gut microbiota analysis
Dynamic changes in the metabolic pathway of gut microbiota between two groups | Day 0.
  Stool sample collection for gut microbiota analysis
Re-infection rate 1 year and 3 years after second line eradication therapy | From Day 0 to Day 56.
  13C-Urea breath tests are performed to check the Helicobacter pylori infection
Changes in the parameters of metabolic syndrome between two groups | Day 0.
  Blood samples are collected for glucose, insulin, HbA1c, and lipid profiles, liver function tests, renal function tests as well as CRP. Also, transabdominal sonography for fatty liver severity assessment would be performed.
Eradication rate of second line BQT between two groups | From Day 0 to 1 year.
  13C-Urea breath tests are performed to check the eradication of Helicobacter pylori between two groups
Eradication rate of second line BQT between two groups | From Day 0 to 3 years.
  13C-Urea breath tests are performed to check the eradication of Helicobacter pylori between two groups
Dynamic changes in the gut microbiota between two groups | Day 10.
  Stool sample collection for gut microbiota analysis
Dynamic changes in the gut microbiota between two groups | Day 56.
  Stool sample collection for gut microbiota analysis
Dynamic changes in the gut microbiota between two groups | 1 year.
  Stool sample collection for gut microbiota analysis
Dynamic changes in the gut microbiota between two groups | 3 years.
  Stool sample collection for gut microbiota analysis
Dynamic changes in the metabolic pathway of gut microbiota between two groups | Day 10.
  Stool sample collection for gut microbiota analysis
Dynamic changes in the metabolic pathway of gut microbiota between two groups | Day 56 .
  Stool sample collection for gut microbiota analysis
Dynamic changes in the metabolic pathway of gut microbiota between two groups | 1 year .
  Stool sample collection for gut microbiota analysis
Dynamic changes in the metabolic pathway of gut microbiota between two groups | 3 years.
  Stool sample collection for gut microbiota analysis
Re-infection rate 1 year and 3 years after second line eradication therapy | From Day 0 to 1 year.
  13C-Urea breath tests are performed to check the Helicobacter pylori infection
Re-infection rate 1 year and 3 years after second line eradication therapy | From Day 0 to 3 years.
  13C-Urea breath tests are performed to check the Helicobacter pylori infection
Changes in the parameters of metabolic syndrome between two groups | Day 56.
  Blood samples are collected for glucose, insulin, HbA1c, and lipid profiles, liver function tests, renal function tests as well as CRP. Also, transabdominal sonography for fatty liver severity assessment would be performed.
Changes in the parameters of metabolic syndrome between two groups | 1 year.
  Blood samples are collected for glucose, insulin, HbA1c, and lipid profiles, liver function tests, renal function tests as well as CRP. Also, transabdominal sonography for fatty liver severity assessment would be performed.
Changes in the parameters of metabolic syndrome between two groups | 3 years.
  Blood samples are collected for glucose, insulin, HbA1c, and lipid profiles, liver function tests, renal function tests as well as CRP. Also, transabdominal sonography for fatty liver severity assessment would be performed.

CONTACTS AND LOCATIONS:
Overall Officials: Ming-Lun Han, doctor, Principal Investigator — National Taiwan University Hospital
Locations (4):
- Taiwan (4):
  - National Taiwan University Hospital Yunlin Branch, Douliu
  - Kaohsiung Medical University Chung-Ho Memorial Hospital, Kaohsiung City
  - National Taiwan University Hospital, Taipei
  - National Taiwan University Cancer Center, Taipei

IPD SHARING:
Plan to Share IPD: No